CLINICAL TRIAL: NCT01303523
Title: Evaluation of the Prevention of Thromboembolic Disease in Patients With a Lower Limb Trauma, Non Surgical, in Winter Sports Resort.
Acronym: M2M-Thrombose
Status: Completed | Type: Observational
Sponsor: Floralis (Industry)
Collaborators: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: DCIC
Record Dates: First submitted 2011-02-23; First posted 2011-02-24 (Estimated); Last update posted 2015-03-06 (Estimated); Status verified 2015-03

CONDITIONS: Leg Injuries; Winter Sport Resorts; Outpatients
Keywords: LMWH; heparin; immobilization; anticoagulant prophylaxis; leg injuries; thromboembolism
MeSH Terms: conditions — Leg Injuries; Thromboembolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to evaluate the impact of thromboembolic diseases and heparin complications in patients with a lower limb trauma supported by physicians of mountain.

DETAILED DESCRIPTION:
The "M2M-thrombose" study is a prospective epidemiological multicenter study involving patients with a lower limb trauma in winter sport resorts. The following initial data required are type of immobilization, treatment with LMWH (Low Molecular Weight Heparin), type of injury (serious or not) and the rolling of the step (normal or abnormal) or no weight bearing.

A 3 month follow-up by phone will be realized by the Investigation Clinical Center in Grenoble. Data about risk factors of thromboembolic diseases, anticoagulant therapy, medical history, new event since inclusion (hospitalization, surgery, lower limb trauma or thromboembolic events) will be collected.

ELIGIBILITY:
Inclusion Criteria:

* patients seen during a consultation with a physician of mountain
* lower limb trauma seen within 48 hours
* patient resident in France

Exclusion Criteria:

* conditions requiring an immediate hospitalization
* prisoners
* pregnant, nursing or parturient woman
* refused participation in follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: outpatients with a lower limb trauma, in winter sports resorts
Sampling Method: Non-Probability Sample
Enrollment: 1627 (Actual)
Dates: Start 2010-12; Primary Completion 2011-03 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
impact of a thromboembolic disease and heparin's complications | 3 months
  Evaluation of the impact of a thromboembolic disease and heparin's complications in outpatients with a lower limb trauma are supported by physicians in winter sports resort. The patients will be contacted by phone 3 months after trauma to collect these data.

SECONDARY OUTCOMES:
compliance with the algorithm for prescribing heparin and consequences on the primary endpoint | 3 months
  The primary endpoint consists to check the impact of thromboembolic disease and adverse effects of anticoagulant therapy at 3 month.
  We compare the link between these consequences and the compliance with the algorithm about the indication of LMWH therapy.
incidence of thromboembolic diseases and heparin complications in different subgroups | 3 months
  Analysis of subgroups depending on the trauma type, the type of immobilization or not, risk factors of thromboembolic diseases, rolling step and weight bearing.
Description of the included patients | evaluation during inclusion visit
  epidemiological description of included patients (age, sex, travel time...)
Epidemiological characteristics of patients with a thromboembolic event or an adverse effect of the treatment | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Dominique LAMY, MD, Principal Investigator — Médecins de Montagne
Locations (28):
- France (28):
  - medical center "Le chevreuil", Autrans
  - Medical center "le pas du lac", Avoriaz
  - Medical center "les Soldanelles", Bellevaux
  - Medical center "le serre d'aigle", Chantemerle
  - Medical center of Combloux, Combloux
  - Medical home, Flaine
  - Medical center of flumet, Flumet
  - Medical Center Brousse, Font-Romeu-Odeillo-Via
  - Medical center of Beauregard - "les cyclamens", La Clusaz
  - Medical group "le Yéti", La Clusaz
  - Medical center, Lanslevillard
  - Medical group "SELARL Sports médecine montagne", Le Grand-Bornand
  - Medical group of Peric, Les Angles
  - Medical center of "Aiguille rouge", Les Arcs
  - Medical center "Val Montjoie", Les Contamines-Montjoie
  - SCP medical "le Bennevy", Les Gets
  - Medical center, Les Orres
  - Medical center, Lullin
  - Medical center of Jaillet, Megève
  - Medical center of Peisey-Vallandry, Peisey Vallandry
  - Resort of Peyragudes, Peyragudes
  - Medical center "le rocher de l'aigle", Saint-François-Longchamp
  - Medical center "Fleur des alpes", Saint-Gervais-les-Bains
  - Medical center, Samoëns
  - Medical center "medival", Val-d'Isère
  - Medical center of Valberg, Valberg Guillaumes
  - Medical center, Vallouise
  - Medical center, Villard-de-Lans

REFERENCES:
- [Background] Motykie GD, Zebala LP, Caprini JA, Lee CE, Arcelus JI, Reyna JJ, Cohen EB. A guide to venous thromboembolism risk factor assessment. J Thromb Thrombolysis. 2000 Apr;9(3):253-62. doi: 10.1023/a:1018770712660. No abstract available. PMID 10728025
- [Background] Edelsberg J, Ollendorf D, Oster G. Venous thromboembolism following major orthopedic surgery: review of epidemiology and economics. Am J Health Syst Pharm. 2001 Nov 1;58 Suppl 2:S4-13. doi: 10.1093/ajhp/58.suppl_2.S4. PMID 11715837
- [Background] Lijfering WM, Rosendaal FR, Cannegieter SC. Risk factors for venous thrombosis - current understanding from an epidemiological point of view. Br J Haematol. 2010 Jun;149(6):824-33. doi: 10.1111/j.1365-2141.2010.08206.x. Epub 2010 Apr 29. PMID 20456358
- [Background] Gensini GF, Prisco D, Falciani M, Comeglio M, Colella A. Identification of candidates for prevention of venous thromboembolism. Semin Thromb Hemost. 1997;23(1):55-67. doi: 10.1055/s-2007-996071. PMID 9156412
- [Background] Eschwege V, Robert A. Strikes in French public transport and resistance to activated protein C. Lancet. 1996 Jan 20;347(8995):206. doi: 10.1016/s0140-6736(96)90393-1. No abstract available. PMID 8544587
- [Background] Vaitkus PT, Leizorovicz A, Goldhaber SZ; PREVENT Investigator Group. Rationale and design of a clinical trial of a low-molecular-weight heparin in preventing clinically important venous thromboembolism in medical patients: the prospective evaluation of dalteparin efficacy for prevention of venous thromboembolism in immobilized patients trial (the PREVENT study). Vasc Med. 2002;7(4):269-73. doi: 10.1191/1358863x02vm449oa. PMID 12710842
- [Background] Cohen AT, Davidson BL, Gallus AS, Lassen MR, Prins MH, Tomkowski W, Turpie AG, Egberts JF, Lensing AW; ARTEMIS Investigators. Efficacy and safety of fondaparinux for the prevention of venous thromboembolism in older acute medical patients: randomised placebo controlled trial. BMJ. 2006 Feb 11;332(7537):325-9. doi: 10.1136/bmj.38733.466748.7C. Epub 2006 Jan 26. PMID 16439370
- [Background] Kujath P, Spannagel U, Habscheid W. Incidence and prophylaxis of deep venous thrombosis in outpatients with injury of the lower limb. Haemostasis. 1993 Mar;23 Suppl 1:20-6. doi: 10.1159/000216905. PMID 8388353
- [Background] Jorgensen PS, Warming T, Hansen K, Paltved C, Vibeke Berg H, Jensen R, Kirchhoff-Jensen R, Kjaer L, Kerbouche N, Leth-Espensen P, Narvestad E, Rasmussen SW, Sloth C, Torholm C, Wille-Jorgensen P. Low molecular weight heparin (Innohep) as thromboprophylaxis in outpatients with a plaster cast: a venografic controlled study. Thromb Res. 2002 Mar 15;105(6):477-80. doi: 10.1016/s0049-3848(02)00059-2. PMID 12091045
- [Background] Lassen MR, Borris LC, Nakov RL. Use of the low-molecular-weight heparin reviparin to prevent deep-vein thrombosis after leg injury requiring immobilization. N Engl J Med. 2002 Sep 5;347(10):726-30. doi: 10.1056/NEJMoa011327. PMID 12213943
- [Background] Riou B, Rothmann C, Lecoules N, Bouvat E, Bosson JL, Ravaud P, Samama CM, Hamadouche M. Incidence and risk factors for venous thromboembolism in patients with nonsurgical isolated lower limb injuries. Am J Emerg Med. 2007 Jun;25(5):502-8. doi: 10.1016/j.ajem.2006.09.012. PMID 17543652